CLINICAL TRIAL: NCT04327869
Title: Feasibility of Using Magnetically-controlled Capsule Endoscopy for Direct Visualization of Drug Behavior in Upper-gastrointestinal Tract
Brief Title: MCE Direct Visualization of Drug Behavior in Upper-gastrointestinal Tract
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, M.D., Associate Professor, Associate Chief Physician, Changhai Hospital
Other Study IDs: MCE_sucralfate gel
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Capsule Endoscopy
Keywords: Magnetically controlled capsule endoscopy; sucralfate gel; drug behavior; upper-gastrointestinal tract
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Abdominal symptoms group: The investigators selected 10 subjects (male: female = 1: 1) from patients with a recent history of upper-gastrointestinal symptoms who met the indication of taking sucralfate suspension gel
  Interventions: Device: Magnetically controlled capsule endoscopy
- Healthy control group: The investigators selected another 10 subjects (male: female = 1: 1) from healthy volunteers.
  Interventions: Device: Magnetically controlled capsule endoscopy

INTERVENTIONS:
Device: Magnetically controlled capsule endoscopy — The subjects swallowed the capsule with water in the left lateral position. When capsule enter stomach cavity, subject was asked to sit up and ingested 4 g aerogenic powder with 5 ml water to distend the stomach, and performed gastric baseline examinations to identify the lesions. After baseline examination, subjects ingested dyed sucralfate gel and performed the first-time examination. The examination was repeated at 30 min intervals, until dyed sucralfate gel disappeared completely.

SUMMARY:
The investigators aim to explore the feasibility of MCE in direct, real-time visualization of drug behavior in upper-gastrointestinal tract, which presented by the adhesion, distribution, and dissipation characteristics of dyed sucralfate gel.

DETAILED DESCRIPTION:
This pilot study was a prospective, single-centered, nonrandomized study. The investigators selected 10 subjects from patients with a recent history of upper-gastrointestinal symptoms who met the indication of taking sucralfate suspension gel, and another 10 subjects from healthy volunteers.

Procedures were performed by the NaviCam magnetic capsule guidance system. To enhance discrimination, the sucralfate gel dyed with 0.3 ml methylene blue. The subjects swallowed the capsule with water in the left lateral position. When capsule enter stomach cavity, subject was asked to sit up and ingested 4 g aerogenic powder with 5 ml water to distend the stomach, and performed gastric baseline examinations to identify the lesions. After baseline examination, subjects ingested dyed sucralfate gel and performed the first-time examination. The examination was repeated at 30 min intervals, until dyed sucralfate gel disappeared completely. When study completed, the capsule was detached from string and continued into the small bowel for further examination.

The endoscopists recorded the adhesion and dissipation times of dyed sucralfate gel, calculated the efficient time, and selected the images of six primary anatomic landmarks from each examination to measure the distribution area (%) . Any complication or discomfort during the procedure was evaluated. The discomfort was scored on a scale from 0 to 3 (0 = no; 1 = mild/minimal; 2 = moderate; 3 = sever/very difficult).

ELIGIBILITY:
Inclusion Criteria:

* With or without gastrointestinal complaints
* Scheduled to undergo a capsule endoscopy for both stomach and small bowel
* Signed the informed consents before joining this study

Exclusion Criteria:

* Suspected or known gastrointestinal stenosis
* Obstruction or other known risk factors for capsule retention
* Pregnancy or suspected pregnancy
* Pacemakers or electromedical devices implanted
* Any other contraindications determined by endoscopists

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers who agreed to participate in the feasibility examination of MCE direct visualization of sucralfate gel behavior in fasted stomach.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-11-03 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Sucralfate gel adhesion behavior in the fasted gastric cavity | 180 minutes
  The adhesion time was recorded from the sucralfate gel entered the stomach to all sucralfate adhered to the gastric wall.
Sucralfate gel distribution behavior in the fasted gastric cavity | 0, 30, 60, 90, 150, 180 min after dyed sucralfate gel enter the stomach
  The distribution area of sucralfate gel was measured by selecting images of six primary anatomic landmarks (cardia, fundus, body, angulus, antrum, and pylorus) at different times, the images were imported into MATLAB software to calculate the area of sucrafate gel. The dynamic changes of distribution area of sucralfate gel over the time were analyzed and performed with GraphPad Prism.
Sucralfate gel dissipation behavior in the fasted gastric cavity | 180 minutes
  The dissipation time was evaluated by calculating the times between sucralfate gel entered the stomach and adhered sucralfate disappeared completely.

SECONDARY OUTCOMES:
Number of Participants with complications of MCE | 2 weeks
  Any complications associated with MCE.
Discomfort scores of participants during the procedure | during the procedure
  The discomfort associated with the procedure included swallow difficulty, nausea caused by string, pulling capsule up and down, abdominal distension or pain caused by ingesting aerogenic powder, discomfort during MCE examination, and pulling the string out. The discomfort was scored on a scale from 0 to 3 (0 = no; 1 = mild/minimal; 2 = moderate; 3 = sever/very difficult).

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, Study Chair — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang YC, Pan J, Jiang B, Qian YY, Qiu XO, Yuan YZ, Li ZS, Liao Z. Direct visualization of drug behaviors in the upper GI tract via magnetically controlled capsule endoscopy. VideoGIE. 2021 May 28;6(7):333-338. doi: 10.1016/j.vgie.2021.04.004. eCollection 2021 Jul. PMID 34278100